CLINICAL TRIAL: NCT07188428
Title: Treatment Patterns and Outcomes Among Patients With Chronic Myeloid Leukemia (CML) in All Lines of Therapy: An Analysis of Medicare Fee-for-Service (FFS) Data
Brief Title: Treatment Patterns and Outcomes Among Patients With Chronic Myeloid Leukemia (CML) in All Lines of Treatment
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001A0US06
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Leukemia, Chronic Myeloid
Keywords: Tyrosine kinase inhibitors; Treatment pattern; Non-optimal treatment profile
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- 1L Cohort: Adult patients newly diagnosed with CML who received 1L treatment with imatinib, dasatinib, nilotinib, or bosutinib.
- 2L Cohort: Adult patients from the 1L Cohort with a subsequent line of treatment (i.e., second treatment) with imatinib, dasatinib, nilotinib, bosutinib, ponatinib, or asciminib.

SUMMARY:
The aim of this study was to evaluate the real-world treatment patterns, healthcare resource use and costs among patients newly diagnosed with CML who were treated with tyrosine kinase inhibitors (TKIs) in first- and second-line therapy.

DETAILED DESCRIPTION:
The study used claims from Medicare FFS data from 1 January 2016 to 31 December 2022 (observation period). The patient identification period spanned from 1 January 2017 to 30 June 2022. The index date was the date of treatment line initiation. Patients were followed from index date until death, end of enrollment, or study end (31 December 2022), whichever came first. Each patient's follow-up was variable in length.

Variables were assessed during the follow-up period in first-line (1L) and second-line (2L) treatment cohorts and were stratified by generations of TKIs and treatment profiles. Patients were categorized into non-optimal treatment (NOPT) profiles and reference groups, and treatment patterns, healthcare resource utilization (HCRU), and payer healthcare costs were summarized descriptively for each group.

ELIGIBILITY:
Inclusion criteria:

1. L Cohort:

   * Patients had at least one diagnosis for CML (International Classification of Diseases, 10th Revision, Clinical Modification [ICD-10-CM]: C92.1x) during the observation period.
   * Patients ≥18 years of age as of the first CML diagnosis.
   * Patients received imatinib, dasatinib, nilotinib, or bosutinib in 1L.
   * Patients initiated 1L within a maximum of 3 months following the first observed CML diagnosis.
   * Patients had at least 12 months of continuous enrollment prior to the index date.
   * Patients had at least 6 months of continuous enrollment post index date (including index date).
2. L Cohort:

   * Patients in the 1L cohort.
   * Patients received imatinib, dasatinib, nilotinib, bosutinib, ponatinib or asciminib in 2L.
   * Patients with at least 12 months of continuous enrollment prior to the index date.
   * Patients with at least 6 months of continuous enrollment post index date (including index date).

Exclusion criteria:

1. L Cohort:

   * Patients with medical services with a procedure code for imatinib any time during the observation period.
   * Patients with a diagnosis for CML remission (identified by ICD-10-CM code: C92.11) or CML relapse (ICD-10-CM code: C92.12) any time in the baseline period before the 1L initiation.
   * Patients with a medical claim associated with a clinical trial drug during the baseline period before the 1L initiation up to the end of the observation period.
   * Patients who received chemotherapy, or a TKI of interest or had a hematopoietic stem cell transplantation (HSCT) during the baseline period before 1L initiation.
2. L Cohort:

   * Patients with a diagnosis for CML remission (identified by ICD-10-CM code: C92.11) or CML relapse (ICD-10-CM code: C92.12) any time before the 2L initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, non-interventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 2298 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Number of Patients Who Switched to Another CML-related Treatment by TKI Generation and Treatment Profile | Up to approximately 6 years
Number of Patients Who Switched to Another CML-related Treatment Within 6 Months of Starting Treatment by TKI Generation and Treatment Profile | 6 months
Time to Treatment Switch by TKI Generation and Treatment Profile | Up to approximately 6 years

SECONDARY OUTCOMES:
Proportion of Days Covered (PDC) by TKI Generation and Treatment Profile | Up to approximately 6 years
  Adherence was assessed using PDC. The PDC was defined as the number of days of medication covered during the treatment line, divided by the number of calendar days between the start and end dates of the line of treatment.
Number of Patients With PDC >80% by TKI Generation and Treatment Profile | Up to approximately 6 years
  Adherence was assessed using PDC. The PDC was defined as the number of days of medication covered during the treatment line, divided by the number of calendar days between the start and end dates of the line of treatment.
Number of Patients who Discontinued Treatment by TKI Generation and Treatment Profile | Up to approximately 6 years
Time to Treatment Discontinuation by TKI Generation and Treatment Profile | Up to approximately 6 years
Number of Patients With Treatment Interruption by TKI Generation and Treatment Profile | Up to approximately 6 years
  Treatment interruption was defined as a gap of ≥14 days in CML treatment with resumption of that treatment after the gap.
Time to First Treatment Interruption by TKI Generation and Treatment Profile | Up to approximately 6 years
Number of Patients With a Dose Reduction by TKI Generation and Treatment Profile | Up to approximately 6 years
Time to Dose Reduction by TKI Generation and Treatment Profile | Up to approximately 6 years
Mean Number of All-cause Healthcare Visits per Person per Year (PPPY) by Treatment Profile | Up to approximately 6 years
  Healthcare visits included inpatient visits, outpatient visits, emergency department visits, and pharmacy visits.
Mean Number of CML-related Healthcare Visits per Person per Year (PPPY) by Treatment Profile | Up to approximately 6 years
  Healthcare visits included inpatient visits, outpatient visits, emergency department visits, and pharmacy visits.
Mean Length of Stay (LoS) of Inpatient Visits PPPY by Treatment Profile | Up to approximately 6 years
Mean All-cause Healthcare Cost PPPY by Treatment Profile | Up to approximately 6 years
  Healthcare costs included:
  * Total costs
  * Inpatient costs
  * Emergency department costs
  * Outpatient costs
  * Other costs
  * Pharmacy costs
Mean CML-related Healthcare Cost PPPY by Treatment Profile | Up to approximately 6 years
  Healthcare costs included:
  * Total costs
  * Inpatient costs
  * Emergency department costs
  * Outpatient costs
  * Other costs
  * Pharmacy costs

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States